CLINICAL TRIAL: NCT06467825
Title: Effect of Sex on Orthostatic Intolerance and Cardiovascular Response During Lunar Descent and Ascent
Acronym: Lunar OI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000460
Record Dates: First submitted 2024-03-07; First posted 2024-06-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Hypovolemic (Experimental): Furosemide and potassium supplement.
  Interventions: Drug: Potassium Supplement; Drug: Furosemide 20 MG
- Hypovolemic plus garment (Experimental): Furosemide and potassium supplement plus OIG.
  Interventions: Drug: Potassium Supplement; Drug: Furosemide 20 MG; Device: Compression Garment

INTERVENTIONS:
Drug: Potassium Supplement — Participants will be given a potassium supplement that will help prevent low blood potassium levels.
  Arms: Hypovolemic; Hypovolemic plus garment
Drug: Furosemide 20 MG — Furosemide (Lasix, 20 mg) will be administered through IV catheter to induce urination. The goal of this procedure is to reduce the volume of plasma in the blood.
  Other Names: Lasix
  Arms: Hypovolemic; Hypovolemic plus garment
Device: Compression Garment — From the torso and leg measurements obtained during Visit 1A, a custom-designed compression garment will be constructed.
  Arms: Hypovolemic plus garment

SUMMARY:
The purpose of Lunar OI (Orthostatic Intolerance) is to determine if there are differences between males and females in tolerance to and cardiovascular responses during different angles of head-up tilt simulating gravity levels less than or equal to Earth's gravity. Also, this study will determine if a gradient compression garment affects tolerance to tilting and the cardiovascular stress at different tilt angles. Males and females are being identified by biological sex. This will be a two-phased study design. In Phase I we will determine whether there are differences in the development of signs or symptoms of orthostatic intolerance between males and females when tilted head up on a table to different angles to simulate gravity levels that astronauts may experience when landing on or launching from the surface of the Moon. In Phase II, the tilt tests simulating the same gravity levels from Phase I will be repeated, but a custom-made lower-body compression garment will be worn to see if wearing the garment affects the development of orthostatic intolerance. For both study phases, before tilting, a drug will be administered to reduce the amount fluid in the blood (plasma) to levels similar to that experienced by astronauts during spaceflight.

DETAILED DESCRIPTION:
Phase I, Visit one Alpha (1A);

OIG (Orthostatic Intolerance Garment) Measurement:

Participants will lie supine while torso and anthropometric measurements are acquired. The investigators will utilize the same procedures developed and adopted by the Orion Program to obtain foot, leg, and torso circumference measurements at pre-determined intervals. This detailed measurement procedure has shown to be effective at providing precise compression levels at pre-determined anatomical locations. The target levels of compression will be verified by the manufacturer, using a Hosiery and Allied Trades Research Association (HATRA) test instrument that is identified in the British Standard for testing compression in elastic stockings.

Tilt Familiarization:

Participants will be instructed to lie supine without moving throughout the Familiarization tilt test. After instrumentation with brachial blood pressure, continuous blood pressure monitoring, and electrocardiogram (ECG) for heart rate, baseline measures will be obtained for at least 2 minutes while the test is explained. Participants will be tilted to 80˚ head-up and instructed to remain still and quiet. After allowing the participant to become familiar with the tilt procedure and the feeling of being upright, the bed will be lowered back to horizontal (flat) and a timer started for a 20-minute supine rest period.

Plasma and Blood Volume Measurement:

An intravenous (IV) catheter will be inserted into a vein in the participant's arm or hand using standard techniques. All blood samples will be obtained using the IV catheter in the participant's arm, unless it becomes clogged, and another IV catheter cannot be placed in another arm or hand vein. In this situation, blood could be drawn from the participant's arm or hand vein using a butterfly needle.

Participants will be supine for 20 minutes before this test begins. A clip will be placed on the participant's nose so that they are breathing only through their mouth. Participants will breathe through a mouthpiece connected to a rebreathing circuit containing 100% oxygen, which is scrubbed by soda lime to remove carbon dioxide. After ~5 minutes, a ~10 mL blood sample will be collected using the IV catheter. Thereafter, a small amount of carbon monoxide will be added into the breathing circuit, and the participant will breathe this mixture of carbon monoxide and oxygen for ~10 min. Then, a second ~10 mL blood sample will be obtained. Analysis of the blood samples (i.e., hematocrit, hemoglobin, and carboxyhemoglobin) will be used to calculate red blood cell mass, plasma volume, and total blood volume.

Normovolemic Tilt Test at one unit of gravity (1G):

This test will be similar to the Tilt Familiarization session, but baseline data will be collected for ~5 minutes while supine. After tilting up, participants will remain quiet, relaxed, and not move for up to 20 minutes or until presyncope. Brachial blood pressure will be measured, and ultrasound images obtained to quantify stroke volume approximately every minute. Blood pressure and ECG will be continuously monitored before, during, and after the tilt. A tilt test will be terminated if any of the following test termination criteria are met: sudden drop in heart rate (>15 bpm), systolic blood pressure (>25 mmHg) or diastolic blood pressure (>15 mmHg); significant cardiac arrhythmias such as an ectopic rhythm >4 beats; absolute systolic blood pressure <70 mmHg; symptoms such as nausea, clammy skin, profuse sweating, pallor, light-headedness, dizziness, or tingling; or participant request. In the event a tilt test is terminated prior to 20 minutes, the participant will be brought to a head-down tilt position until recovered.

Visit one Bravo (1B);

Plasma Volume + Furosemide Infusion:

Plasma volume will be measured as described in Phase 1A. After the plasma volume test is complete, a 20 mg of Furosemide will be administered intravenously. This dose has been demonstrated to produce plasma volume losses similar to spaceflight and bedrest. An oral potassium supplement of 20 mEq (Milliequivalent) will be given as a prophylactic prior to the furosemide infusion.

Induction of Hypovolemia:

Following Furosemide infusion, participants will remain in the CVL (Cardiovascular and Vision Laboratory) and be observed while remaining seated (except for bathroom trips) for 2 hours. During this time urine volume and periodic blood pressure will be obtained. Participants will self-collect urine using urine collection bottles and provide to the test operator to document the time of urine collection and volume produced. Participants will be given a standardized volume of water at intervals throughout the study day. Participants will be provided snacks as needed throughout the duration of their stay in the laboratory.

Hypovolemic Tilt Tests (1-G, 0.75-G, 0.50-G):

Following the 2-hour period for diuresis to develop, participants will undergo 3 tilt tests (80°, 50°, and 30° head-up tilt) for up to 20 minutes each to simulate 1-G, 0.75-G, and 0.50-G exposures. The tilt tests will occur in a random order and participants will remain supine for 20 minutes to fully recover between tests. The timing, monitoring, and test termination criteria will be identical to that described in Normovolemic Tilt Test (1G) above. Immediately prior to each tilt test, a blood sample (5 mL) will be drawn using the IV catheter and analyzed for hematocrit and hemoglobin concentration, which will then be used to calculate the change in plasma volume since the baseline test. Alternatively, if the IV becomes clogged and another IV cannot be placed, these blood samples could be drawn from an arm or hand vein using a butterfly needle (5 mL) or by pricking the finger (80 μL).

Phase II, Visit two Alpha (2A);

OIG Fit Check:

Participants will don their custom OIG garments to ensure there were no errors in garment development.

Visit two Bravo (2B):

Plasma Volume + Furosemide Infusion Participants will complete the same testing protocol as occurred in Phase 1B.

Induction of Hypovolemia:

Participants will complete the same testing protocol as occurred in Phase 1B.

Hypovolemic Tilt Tests (1-G, 0.75-G, 0.50-G) + OIG:

Following the 2-hour period for diuresis to develop, participants will don their custom-made OIG and assume the supine posture for ~20 minutes prior to starting the first tilt test. The order of the 3 tilt tests (80°, 50°, and 30° head-up tilt) will be the same order as occurred in Phase 1B, Hypovolemic Tilt Tests (1-g, 0.75-G, 0.50-G).

Visits 2A and 2B can be combined.

ELIGIBILITY:
Inclusion Criteria:

• Pass a test subject screening facility modified Air Force Class III physical

Exclusion Criteria:

* Known allergy to furosemide or sulfa drugs
* Currently taking drugs or medications known to adversely interact with furosemide, including but not limited to aspirin, NSAIDs, antibiotics, or immunosuppressant drugs
* Systemic diseases or current medications known to influence the cardiovascular system
* Renal disease
* Type II Diabetes
* Pregnant participants will be excluded (a urine pregnancy screen will be made available).

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Plasma Volume | 7-8 hours
  Plasma volume and change in plasma volume is calculated using the Dill and Costill equation cited here: Dill DB, Costill DL. Calculation of percentage changes in volumes of blood, plasma, and red cells in dehydration.
Tilt Tolerance Time | 0-20 minutes
  duration of Tilt Test
Heart Rate | 0-20 minutes
  beats per minute
Blood Pressure | 0-20 minutes
  systolic and diastolic, continuous blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- NASA, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No